CLINICAL TRIAL: NCT07277530
Title: A Nurse-Led Nutritional Education Intervention Reduces Serum Potassium in Moroccan Hemodialysis Patients Lacking Dietitian Support.
Brief Title: Nurse-Led Nutritional Education for Moroccan Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HASSAN 1st university (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERS/UEMF-2025/EC10/02; CERS/UEMF-2025/EC10/02 (Other: Euro-Mediterranean University of Fez Ethics Committee)
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease 5D; Hyperkalemia; Hemodialysis
Keywords: Hemodialysis; Nurse-Led; Nutritional Education; Hyperkalemia Management; Interdialytic Weight Gain; Quality of Life
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Intervention Model Description: This is a pre-post experimental investigation. All participants were assigned to the single intervention group and acted as their own controls, with outcomes measured before (T0) and after (T1) the nurse-led nutritional education program. There was no separate control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Education Intervention (Experimental): This arm represents the single group in this pre-post study. All 30 participants received the educational intervention over five months (Feb-June 2025). The program focused on dietary management of potassium and fluid, salt intake, and physical stretching exercises, delivered by a nurse in the Moroccan dialect.
  Interventions: Behavioral: Nutritional Education Intervention

INTERVENTIONS:
Behavioral: Nutritional Education Intervention — Educational sessions focused on dietary management of potassium and fluid restriction, salt intake, and low-impact physical activity (stretching). The program was delivered by a nurse in the Moroccan dialect via face-to-face and remote (WhatsApp) communication.

SUMMARY:
Why was this study done? Many dialysis centers in Morocco lack dietitians to provide proper, individualized dietary support to patients. High potassium levels (hyperkalemia) are a major risk factor for heart problems in dialysis patients. This study tested whether a simple nutritional education program, led by a nurse, could help patients better manage their diet and safely reduce their serum potassium levels.

Who participated? Thirty (30) adult patients with end-stage renal disease receiving hemodialysis participated in the study. They were recruited from three public hemodialysis centers in Morocco that did not have permanent dietitians.

What did participants do? The study was conducted from February to June 2025. Participants received an educational intervention led by a nurse. The sessions covered potassium content in food, fluid intake, thirst management, and physical activity.

What did the study find (Results)? The educational program resulted in a statistically significant reduction in patients' serum potassium levels. The percentage of patients within the ideal potassium range (4 to 5 mmol/L) increased from 36.7% at the start to 46.7% at the end. This demonstrates that a nurse-led program is a practical and beneficial approach to help lower cardiovascular risk in resource-scarce settings.

The study found no significant changes in Quality of Life (QoL) or interdialytic weight gain (IDWG).

DETAILED DESCRIPTION:
This is a single-group, pre-post interventional study designed to evaluate the impact of a nurse-led nutritional education program on the management of End-Stage Renal Disease (ESRD) patients undergoing hemodialysis in a resource-limited setting in Morocco. The study enrolled 30 adult patients.

The intervention was conducted over five months (February to June 2025). The program was delivered by a nurse and included face-to-face sessions as well as remote support (WhatsApp). The educational content focused on three main areas:

Dietary management to reduce hyperkalemia (potassium content in food). Fluid restriction and thirst management. Salt restriction and low-impact physical activity. The primary outcome measure was the change in serum potassium levels (Kalemia) from baseline (T0) to post-intervention (T1). Secondary outcomes included changes in interdialytic weight gain (IDWG) and Quality of Life (QoL).

The results demonstrated a statistically significant reduction in patients' serum potassium levels, supporting the practical benefits of the nurse-led program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease (ESRD) undergoing maintenance hemodialysis. Participants must have provided written informed consent.

Exclusion Criteria:

* Patients who declined to participate; patients who were minors (under 18 years old); and patients with conditions impairing their ability to understand or receive educational content, such as severe hearing loss or cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Serum Potassium Level | From baseline to 12 weeks after the start of the intervention.
  Change in serum potassium concentration measured at baseline (T0) and after the 12-week educational intervention (T1).

SECONDARY OUTCOMES:
Change in Interdialytic Weight Gain (IDWG) | 4 weeks before baseline and 4 weeks at the end of the 12-week intervention
  Change in interdialytic weight gain, calculated as the mean IDWG during the 4 weeks before baseline and the 4 weeks at the end of the 12-week educational intervention
Change in Quality of Life (QoL) Index Score | From baseline to 12 weeks after the start of the intervention.
  Measured using the validated Arabic version of the EuroQol 5 Dimensions (EQ-5D-5L) instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Settat Hemodialysis Center,el borouj Hemodialysis Center, Al amal Hemodialysis Center, Settat, Settat, Morocco

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article (e.g., serum potassium levels, IDWG, and EQ-5D-5L scores) will be shared. Data will be made available upon request to the Principal Investigator (PI), following the publication of the final article. The data will be de-identified to protect participant privacy. Requests should be justified and may require an institutional agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be available starting six months after publication of the final article and will remain available for a period of five years (until 2030).
Access Criteria: The identified individual participant data (IPD) and supporting documentation will be accessible to qualified researchers who submit a methodologically sound and ethically approved proposal to the Principal Investigator (PI). Access will be granted via a secure shared drive after signing a data access agreement.
URL: https://ueuromed.org/innovation/research-project